CLINICAL TRIAL: NCT01220154
Title: Phase I Study of Intraperitoneal Carboplatin With Intravenous Paclitaxel and Bevacizumab in Patients With Previously Untreated Epithelial Ovarian Carcinoma or Primary Peritoneal Carcinoma
Brief Title: Study of Intraperitoneal Carboplatin With IV Paclitaxel and Bevacizumab in Untreated Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David O'Malley (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David O'Malley, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09115; NCI-2012-00341 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2025-02-21 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; No Prior Chemotherapy
Keywords: ovarian; cancer; fallopian tube; peritoneal; intraperitoneal; bevacizumab; carboplatin; paclitaxel; chemo-naive
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin Paclitaxel & Bevacizumab (Experimental): Intraperitoneal carboplatin with weekly intravenous paclitaxel and intravenous bevacizumab
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — Cycle 1 Day 1, 8, 15 IV 60-80mg mg/m2 as a 1 hour infusion. For cycle 2-6 Day 1,8,15 IV 60-80 mg/m2 as 1 hour infusion. Repeat every 3 weeks times 5 cycles.
  Other Names: Abraxane; Taxol
Drug: Carboplatin — Intraperitoneal Day 1 cycles 1-6 AUC
  Other Names: Paraplatin®
Drug: Bevacizumab — Bevacizumab 15 mg/kg intravenous infusion Day 1 cycles 2-6 Optional cycles 7-22 15 mg/kg intravenous infusion Day 1 every 21 days
  Other Names: Avastin

SUMMARY:
Phase I study to evaluate intraperitoneal carboplatin along with weekly intravenous paclitaxel and bevacizumab in order to establish a tolerable dose and define the toxicity of this regimen in previously untreated patients with advanced ovarian carcinoma.

DETAILED DESCRIPTION:
Phase I study with the primary objective to determine the maximum tolerated dose of intraperitoneal carboplatin and intravenous weekly paclitaxel given in combination with intravenous bevacizumab during the second two cycles of treatment in patients with chemo-naive epithelial ovarian, primary peritoneal or fallopian tube cancer. The maximum tolerated dose is defined as the highest dose at which no more than 1 of 6 evaluable patients experiences a dose limiting toxicity during the second two cycles of treatment. Secondary objectives are to determine response rates and to estimate progression free survival and overall survival of this class of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histology diagnoses epithelial ovarian, primary peritoneal, or fallopian tube(Stage II, III or IV)either optimal or suboptimal after initial surgery.

  * All patients must have had appropriate surgery for ovarian, peritoneal, or fallopian tube carcinoma with tissue available for histologic evaluation
  * Histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant brenner tumor, adenocarcinoma NOS.
* GOG(Gynecologic Oncology Group)performance status of 0,1,2
* Entered within 12 weeks of most recent surgery performed for diagnosis.
* Patients must have adequate bone marrow function, renal function,hepatic function, neurologic function, blood coagulation parameters within normal limits
* Sign approved consent form.

Exclusion Criteria:

* Patients who have received prior treatment other than initial surgery
* Patients who have received prior radiotherapy to any portion of their abdominal cavity or pelvis
* Patients with acute hepatitis or active infection
* Patients with active bleeding
* Patients with unstable angina
* Patients with history of invasive malignancies with the exception of nonmelanoma skin cancer and localized breast cancer.
* Patients who have received any target therapy or hormonal therapy for management of their ovarian cancer.
* Patients with synchronous primary endometrial cancer.
* Patients with epithelial tumors of low malignant potential
* Serious non healing wound, ulcer or bone fracture.
* Patients with history or evidence of CNS(central nervous system disease)
* Patients under 18 years old.
* Patients who have received prior therapy with anti-VEGF(vascular endothelial growth factor)

drug, bevacizumab

* Patients who have a history of allergic reaction to polysorbate 80.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Every Cycle-28 days
  The Maximum Tolerated Dose is defined as the highest dose at which no more than 1 of 6 evaluable patients experiences a dose limiting toxicity.

SECONDARY OUTCOMES:
Response Rate, Progression Free Survival and Overall Survival | Every 3 monthes for 2 years, Every 6 months for 3 years.
  Response Rate in patients with measurable disease using the RECIST(Response Evaluation Criteria in Solid Tumors)criteria.
  Progression free survival is also uses the RECIST criteria or GCIG criteria. Overall survival will be followed for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: David O'Malley, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- OSU Gyn Oncology at Mill Run, Hilliard, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu